CLINICAL TRIAL: NCT06078358
Title: The Effects of Resistance Exercise on Muscle Activation and Lipids in Children
Brief Title: Resistance Exercise Training in Children.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Strength and Conditioning Association (Other)
Responsible Party: Principal Investigator, Trent J. Herda, Ph.D., Professor, University of Kansas Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00147248
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Resistance Training
Keywords: exercise; muscle cross-sectional area; intramyocellular lipids; extramyocellular lipids; strength
MeSH Terms: conditions — Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance exercise training (Experimental): Participants undergo 8 weeks (3 days/week) of resistance exercise training.
  Interventions: Other: Resistance exercise training
- Control (No Intervention): Participants do not perform 8 weeks of resistance exercise training.

INTERVENTIONS:
Other: Resistance exercise training — Traditional linear periodization resistance training.
  Arms: Resistance exercise training

SUMMARY:
The purpose of this study is examine the effects of 8 weeks (3 days/week) of resistance exercise training in children 8 to 10 years of age on muscle strength, activation, and lipids of the vastus lateralis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer males and females ages 8 - 10 years.

Exclusion Criteria:

* No history or ongoing neuromuscular diseases, musculoskeletal injuries, or a disease that effects metabolism.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-09-06 (Actual)

PRIMARY OUTCOMES:
Change in the muscular strength of leg extensors, as measured with isometric strength. | baseline, following the intervention (9 weeks)
  The score will reflect the strength of the leg extensors. The higher score, reflects greater muscular strength.

SECONDARY OUTCOMES:
Change from baseline in motor unit firing rates during a 60% of maximal voluntary contraction (MVC). | baseline, following the intervention (9 weeks)
  Scores are measured with the y-intercept from the firing rates versus recruitment threshold relationships from the 60%. The higher y-intercept score reflects greater muscle activation.
Change from baseline in motor unit firing rates during a 60% of maximal voluntary contraction (MVC). | baseline, following the intervention (9 weeks)
  Scores are measured with the slope from the firing rates versus recruitment threshold relationships from the 60%. The higher slope score reflects greater muscle activation.
Change from baseline in thigh muscle cross-sectional area. | baseline, following the intervention (9 weeks)
  Scores are measured cross-sectional area from ultrasound images.

OTHER OUTCOMES:
Change from baseline in the fatty acid saturation levels of the extramyocellular lipids of the vastus lateralis, as measure with magnetic resonance spectroscopy | baseline, following the intervention (9 weeks)
  The score will reflect a saturation level of fatty acids in the extramyocellular lipid. The higher score, reflects greater fatty acid saturation.
Change from baseline in the fatty acid saturation levels of the intramyocellular lipids of the vastus lateralis, as measure with magnetic resonance spectroscopy | baseline, following the intervention (9 weeks)
  The score will reflect a saturation level of fatty acids in the intramyocellular lipid. The higher score, reflects greater fatty acid saturation.
Change from baseline in motor unit firing rates during a 35% of maximal voluntary contraction (MVC). | baseline, following the intervention (9 weeks)
  Scores are measured with the y-intercepts from the firing rates versus recruitment threshold relationships from the 35%. The higher y-intercept score reflects greater muscle activation.
Change from baseline in motor unit firing rates during a 35% of maximal voluntary contraction (MVC). | baseline, following the intervention (9 weeks)
  Scores are measured with the slopes from the firing rates versus recruitment threshold relationships from the 35%. The higher slope score reflects greater muscle activation.
Change from baseline in intramyocellular lipids of the vastus lateralis, as measure with magnetic resonance spectroscopy | baseline, following the intervention (9 weeks)
  The score will reflect a concentration. The higher score, reflects more fat in the fibers.
Change from baseline in extramyocellular lipids of the vastus lateralis, as measure with magnetic resonance spectroscopy | baseline, following the intervention (9 weeks)
  The score will reflect a concentration. The higher score, reflects more fat in the fibers.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Hoglund Biomedical Imaging Center, Kansas City, Kansas
  - Exercise and Human Performance Laboratory, Overland Park, Kansas
  - Metabolic and Body Composition Laboratory, Overland Park, Kansas
  - Energy Balance Laboratory, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF